CLINICAL TRIAL: NCT06299813
Title: A Double-blind, Placebo-controlled Randomized Study Comparing the Effectiveness of a Single Dose of Betamethasone vs Placebo in Children With Symptomatic Adenovirus Infection
Brief Title: Effectiveness of a Single Dose of Betamethasone in Children With Symptomatic Adenovirus Infection
Acronym: Adeno-beta
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Claudia Bondone, medical doctor, chief of Department of Pediatric Emergency, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 771.284; 2022-002955-20 (EudraCT Number)
Record Dates: First submitted 2023-12-06; First posted 2024-03-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Adenovirus
Keywords: children; adenovirus; fever; betamethasone
MeSH Terms: conditions — Adenoviridae Infections; Fever | interventions — betamethasone sodium phosphate; Betamethasone

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The nurse that will prepare and administer the treatment to the patient won't be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bentelan (Experimental): The experimental treatment will consist of the active ingredient betamethasone, specifically using the medication Bentelan 0.5mg® effervescent tablets. A single dose of betamethasone will be administered according to the weight categories (0.5 mg if the patient's weight is greater than 5 and less than or equal to 7; 1 mg if the patient's weight is greater than 7 and less than or equal to 12; 1.5mg if the patient's weight is greater than 12 and less than or equal to 17; 2.0 mg if the patient's weight is greater than 17 and less than or equal to 22; 2.5 mg if the patient's weight is greater than 22 and less than or equal to 27.)
  Interventions: Drug: Bentelan
- Placebo (Placebo Comparator): The placebo used in the study will consist of 100 ml of purified water (PPI BBU). The water will be administered in an identical manner to the medication and, like the medication, will be odorless, tasteless, and visually indistinguishable, making it unrecognizable to parents. Regarding the patient population, the study population will primarily consist of infants and preschool-aged children, an age group where the palatability of the medication is perceived to be similar to that of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bentelan — The experimental treatment group will be administered betamethasone 0.1 mg per kg.
  Other Names: Betamethasone
  Arms: Bentelan
Drug: Placebo — The placebo used in the study will consist of 100 ml of purified water (PPI BBU).
  Arms: Placebo

SUMMARY:
The goal of this double-blind, Placebo-controlled Randomized Study is to assess if a single dose of betamethasone in children with febrile adenoviral infection works well in achieving an early fever regulation.

The experimentation is conducted to answer this question: "Can betamethasone help reduce fever more quickly in a child with viral adenovirus infection? "The secondary objective is to assess if the child's overall clinical conditions improve more rapidly (reduced sore throat, quicker return to regular eating) and a reduction in the incidence and duration of hospitalizations.

DETAILED DESCRIPTION:
Adenovirus pharyngitis is a highly febrile illness and tends to last for up to 5-7 days if treated only with antipyretics. Currently, there are no evidence-based effective treatments for this infection. The use of single-dose betamethasone is believed to be effective in significantly reducing the hyper-inflammation that the virus can induce in pediatric patients. However, it is an empirical therapeutic practice used variably because positive clinical experience encourages its prescription but lacks experimental evidence.

The main question at hand is whether the single administration of betamethasone at a dosage of 0.1 mg/kg is truly effective in symptomatic adenoviral infection and whether it can, therefore, reduce the overall fever duration and improve the clinical condition of the children. The study does not involve changes to current clinical practice but aims to demonstrate that this clinical practice, mostly used empirically, is actually based on scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

* Body Temperature measured with an axillary or ear thermometer >= n 37.5°C, persisting for a minimum of 6 hours and a maximum of 5 days.
* Clinical presentation consistent with pharyngo-tonsillar infection by Adenovirus, including At least one of the following symptoms: pharyngodonidae /asthenia/nausea/vomiting/diarrhea/cough/rhinorrhea/abdominal pain/otalgia and at least one of the following signs: pharyngeal hyperemia with or without pharyngo-tonsillar exudate/inflammation of the upper or lower airways/lymphadenopathy/skin rash.-
* Positive result on the antigen test for Adenovirus performed with the "Biosensor" rapid swab.
* Negative result on the swab for Group A Streptococcus (SBEGA), if deemed necessary following McIsaac criteria
* Informed consent form for participation in the study signed by the parent(s) or legal guardian.

Exclusion Criteria:

* Adequate dosage of betamethasone in the 48 hours prior.
* Underlying chronic illness associated with an increased risk of unusual or severe adenoviral infection.
* Inability to tolerate oral medications.
* Documented allergy or any other known contraindication to Bentelan 0.5mg® medication.-Patients on chronic therapy with anticholinesterases, salicylates, nonsteroidal anti-inflammatory drugs, thiazides, furosemide, amphotericin, xanthines (theophylline), antidiabetic drugs, insulin, cyclosporine, ritonavir, ketoconazole, acetylsalicylic acid, phenytoin, phenobarbital, ephedrine, rifampicin, anticoagulants.
* Subacute or chronic conditions requiring a higher equivalent dose of betamethasone or known primary or secondary adrenal insufficiency.
* Transfer to another hospital for any reason.
* Parents who are unable to understand the proposed study or cannot reliably participate in phone follow-up due to significant language barriers.
* Participation in another study involving an experimental drug within the 30 days prior to and during the current study.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a sustained fever resolution at 24 hours from randomization | at 18 and 24 hours from randomization
  The proportion of patients achieving sustained fever resolution at 24 hours from is the proportion of patients with a a body temperature <37.5°C at 18 and 24 hours from randomization.

SECONDARY OUTCOMES:
Pharyngeal-tonsillar pain level in patients younger than 36 months | from the date of randomization, up to 72 hours
  According to the patient age, the pharyngeal-tonsillar pain level of the child will be measured by the FLACC (Face, Legs, Activity, Cry, Consolability) scale in patients younger than 36 months.
  FLACC mean value 5 points on ten.
Hospitalization | from date of randomization until the date of discharge from emergency department, up to 72 hours
  The proportion of patients admitted following emergency access.
Duration of hospitalization (among those hospitalized), measured in days | from date of randomization until the date of discharge,up to 72 hours
  Number of days from admission date to discharge date.
Cumulative incidence of fever resolution | from date of randomization to 72 hours from randomization
  Cumulative incidence of fever resolution is measured from randomization until the fever resolution confirmed by measurement at the subsequent timepoint; patients without fever resolution within the time of the last fever assessment are censored at this time.
Fever duration | from date of randomization until 72 hours from randomization
  Time from randomization until the first measurement with Body Temperature<37.5°C
Pharyngeal-tonsillar pain level in patients older than 36 months | from the date of randomization, up to 72 hours
  According to the patient's age, the pharyngeal-tonsillar pain level of the child was measured by the Faces Pain Rating Scale (Wong-Baker Scale) in patients with age more or equal to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bondone, MD, Principal Investigator — AOU Città della Salute e della Scienza
Locations (1):
- Ospedale Infantile Regina Margherita, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data requests should be submitted to the corresponding author for consideration. Access to deidentified participant data may be granted following review, after the publication of major results
Supporting Information: Study Protocol
Time Frame: Data will be available after 6 months from major results publication and for the following 5 years
Access Criteria: Data requests should be submitted to the corresponding author for consideration.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT06299813/Prot_SAP_000.pdf